CLINICAL TRIAL: NCT03191032
Title: Cortical and Functional Responses to an Early Protocol of Sensory Re-education of the Hand Using Audio-tactile Interaction
Brief Title: Early Sensory Re-education of the Hand With a Sensor Glove Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Fundação de Apoio ao Ensino, Pesquisa e Assistência do Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto da Universidade de São Paulo (Other)
Responsible Party: Principal Investigator, Marisa de Cassia Registro Fonseca, Collaborator, University of Sao Paulo
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Sensor glove
Record Dates: First submitted 2017-06-02; First posted 2017-06-19 (Actual); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: Peripheral Nerve Injuries
Keywords: Peripheral nerves/lesions; hands; rehabilitation; fMRI
MeSH Terms: conditions — Peripheral Nerve Injuries | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training Group (Experimental): Early sensory re-education of the hand protocol with a sensor glove model, after a median and/or ulnar nerve injury repair
  Interventions: Other: Early sensory re-education of the hand with a sensor glove model
- Control Group (No Intervention): Conventional rehabilitation for peripheral nerve injuries if the hand, without application of any kind of early sensory re-education protocol

INTERVENTIONS:
Other: Early sensory re-education of the hand with a sensor glove model — Training Group patients were submitted to application of a three-month protocol for early sensory re-education of the hand using the sensor glove model developed by Mendes et al. (2011). Patients also received conventional physical therapy for this type of injury in a specialized hand therapy center in a university hospital. Control Group patients received only conventional physical therapy treatment. No home sensory re-education program was established for any group and the CG patients were not submitted to any protocol for early sensory re-education of the hand.
  Other Names: Physical Therapy
  Arms: Training Group

SUMMARY:
The implementation of early sensory re-education (SR) techniques, aimed to preserve the cortical hand area, such as the use of audio-tactile interaction, becomes an important strategy to obtain also a better sensory function. The aim of this study was to investigate sensory function outcomes (threshold monofilaments, two-point discrimination test, STI and DASH) and cortical responses (fMRI) in patients submitted to an early protocol of SR of the hand with a sensor glove model. After surgical repair of median and/or ulnar nerves, 17 participants were divided into two groups: the training group, trained on the protocol with the sensor glove model, and the control group, untrained. After six-month follow-up, no difference was observed between groups, related to sensory function, especially tactile gnosis. Despite this, the early training with this sensor glove model seems to provide some type of cortical audio-tactile interaction, contributing to previous studies that focus in early SR of the hand using the integration of different sensory modalities.

ELIGIBILITY:
Inclusion Criteria:

- Injury of the ulnar and/or median nerves at the wrist or distal forearm level surgically repaired

Exclusion Criteria:

* Neurological diseases
* Systemic diseases, which affected either directly or indirectly the central or peripheral nervous system
* Extensive traumas in the upper limbs

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2014-03 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Sensory Threshold - Mann Whitney non-parametric test | First, Third and Sixth month post-operative
  Sensory Threshold was assessed by esthesiometry at first, third and sixth month post-operative
Tactil Gnosis - Mann Whitney non-parametric test | First, Third and Sixth month post-operative
  Tactile Gnosis was assessed by Two-point discrimination and Shape and Texture Identification Test at first, third and sixth month post-operative
Self-report function - Mann Whitney non-parametric test | First, Third and Sixth month post-operative
  Self-report function was assessed by DASH questionnaire at first, third and sixth month post-operative
Cortical responses - fMRI data analysed by Granger Causality Map | Three months
  Training group subjects were submitted to fMRI exam at third month post-operative

CONTACTS AND LOCATIONS:
Overall Officials: Raquel M Sugano, PhD, Principal Investigator — University of Sao Paolo

IPD SHARING:
Plan to Share IPD: No